CLINICAL TRIAL: NCT03626974
Title: The Calming Effect of Vanilla Odor on Preterm Infant Without Mother's Breast Milk Feeding
Acronym: VANILLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator is gone
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-10; 2017-A00496-47 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth | interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venipuncture with vanilla odor (Experimental): the venipuncture will be performed on the neonate in the presence of a diffuser spreading the vanilla odor and ingestion of water
  Interventions: Biological: Venipuncture; Device: Diffuser spreading odor
- Venipuncture without odor (Placebo Comparator): the venipuncture will be performed with an odorless diffuser and ingestion of sucrose
  Interventions: Biological: Venipuncture; Device: Diffuser spreading odor

INTERVENTIONS:
Biological: Venipuncture — Venipuncture for blood collection
Device: Diffuser spreading odor — Diffuser will place under a Hood with an air-flow

SUMMARY:
Pain is a frequent occurrence during the early life of premature newborns. Studies on the short term effects of pain, and potential for long-term ones, have shown that pain affects various physiological and behaviorial parameters. Sucrose during a painful procedure reduce behaviorial and cardiac manifestations in preterm infant, but a recent study casts doubt on its efficacy. Analgesic treatments are available, but a large number of experimental studies in animals ended up with questioning the safety of their use in neonates, particularly in premature ones. Soothing and analgesic methods have been developed such nonnutritive suckling, sucrose, skin to skin contact, and breastfeeding. Therefore, it is important to explore other methods of analgesia. Recently, the role of olfaction as a soothing tool in full term newborns was examined in several studies. The olfactory system is more mature at birth than the others senses. The neonates reacted with significant facial and respiratory changes to low concentration of olfactory stimuli during the various behaviorial states. The analysis of olfacto-facial configurations revealed that behaviorial markers of disgust discriminated between some odors judged as pleasant and unpleasant by adults rather.

Objective The study was designed to assess the analgesic effect of vanilla odor on preterm neonates. The primary outcome was the Premature Infant Pain Profile (PIPP) score. The secondary outcomes were: the French scale Faceless Acute Neonatal pain Scale (FANS), salivary cortisol.

Study design This is a prospective, randomized, controlled, double-blind and monocentric trial. It is conducted in a level III maternity unit at the North Hospital in Marseille. The infant will feed without their own mother's breast milk, clinically stable, born between 30 and 36 weeks and 6 days gestational age, and of less than 10 days postnatal age. In both groups, the painful stimulus is a venipuncture for blood collection. In the experimental group, called "vanilla odor" group, the venipuncture will be performed on the neonate in the presence of a diffuser spreading the vanilla odor and ingestion of water. In the control group, the venipuncture will be performed with an odorless diffuser and ingestion of sucrose. Both group have non nutritive sucking. The diffuser will place under a Hood with an air-flow of 7 l/min. It will manually switch on 3 minutes before the venipuncture and switch off 3 minutes later. The type and quantity of vanillin to be used were determined during a pre-testing phase. Assessment Scale shows significant improvement in the neonates, with good interobserver agreement.

Attempt results A current randomized study compare effects of breast milk and vanilla odors, on premature neonate's pain during and after venipuncture. Our previous study has shown that maternal breast milk odor in preterm neonates reduces PIPP scores during a venipuncture and markedly reduces crying after this procedure. Therefore, from a clinical perspective, the odor of mother's own breast milk has an analgesic effect on the premature neonate. Olfactory stimulation using maternal breast milk odor could have other clinical implications in neonatal medicine in addition to pain prevention, as does olfactory stimulation with a pleasant vanilla-based odor. It could be integrated into developmental care of premature neonates.

ELIGIBILITY:
Inclusion Criteria:

* Nourished with donated or artificial breast milk
* Term of the certain child
* Child whose post-natal age is less than or equal to 10 days at the time of inclusion
* Eutrophic child
* Child of a non-diabetic mother
* Clinically stable child
* Stop Control Positive Airway Pressure (CPAP) nasal for 48 hours.
* No analgesic or sedative drugs since birth
* Child not presenting a gene syndrome, a progressive neurological disease, a malformative pathology, a cleft lip and palate
* Child whose two parents or legal representatives have accepted their child's participation in this study, and have signed informed consent.

Exclusion Criteria:

* Hypotrophic child greater than 5th percentile on the curves
* Milk-fed child of a mother born to her own mother
* Child over the age of 10 days
* Child with grade 3-4 intraventricular hemorrhage, periventricular leukomalacia, or ulcerative necrotizing enterocolitis

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2023-05-07 (Actual)

PRIMARY OUTCOMES:
the Premature Infant Pain Profile (PIPP) score. | 36 months
  Expression of behavioral signs after the venipuncture. 7 items including 3 behavioral, 2 physiological and 2 contextual, for a score from 0 to 21 depending on the term of the child. A score of at least 6 indicates a painful condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — ASSISTANCE PUBLIQUE HÔPITAUX MARSEILLE
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided